CLINICAL TRIAL: NCT01040832
Title: A Phase II, Open-label, 1:1 Randomized, Controlled Trial Exploring the Efficacy of EMD 1201081 in Combination With Cetuximab in Second-Line Cetuximab-Naïve Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (R/M SCCHN)
Brief Title: EMD 1201081 in Combination With Cetuximab in Second-Line Cetuximab-Naïve Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200068-006
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2014-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck Cancer
Keywords: Head and Neck Cancer; Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Cancer; Cetuximab; EMD 1201081
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Cetuximab; IMO-2055

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab plus EMD 1201081 (Experimental)
  Interventions: Drug: Cetuximab; Drug: EMD 1201081
- Cetuximab monotherapy (Active Comparator)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab weekly (initial dose 400 milligram per square meter [mg/m^2] over 120 minutes followed by 250 mg/m^2 intravenous infusion over 60 minutes) will be administered in 3-week treatment cycle until disease progression. The total treatment period will be approximately 18 months.
  Other Names: Erbitux®
Drug: EMD 1201081 — EMD 1201081 weekly (0.32 milligram per kilogram [mg/kg] by subcutaneous injection) will be administered in 3-week treatment cycle until disease progression. Subjects who will discontinue cetuximab due to toxicity in cetuximab monotherapy, could continue to receive EMD 1201081 monotherapy until disease progression. The total treatment period will be approximately 18 months.
  Other Names: IMO-2055
  Arms: Cetuximab plus EMD 1201081

SUMMARY:
The purpose of this study is to determine if EMD 1201081 in combination with cetuximab is more efficient than cetuximab alone to control the cancer.

EMD 1201081 is an immune modulatory oligonucleotide (IMO) containing phosphorothioate oligodeoxynucleotide and acts as an agonist of Toll-like receptor 9 (TLR9).

EMD 1201081 has been studied in six clinical trials in over 170 subjects either as a monotherapy or in combination with chemotherapeutic agents or targeted therapies. Two studies have been conducted in healthy volunteers. In the other five studies, subjects with advanced solid tumors, renal cell carcinoma, non-small cell lung cancer and colorectal cancer have been treated with EMD 1201081. Two studies are still ongoing. Future clinical development of EMD 1201081 will focus on colorectal cancer (CRC) and squamous cell cancer of the head and neck (SCCHN).

In this Phase 2 study, subjects with recurrent or metastatic squamous cell cancer of the head and neck (R/M SCCHN), will be treated with cetuximab plus EMD 1201081 or cetuximab alone. The study will be conducted as a multicenter study in several European Union (EU) member states and the Unites States.

EMD 1201081 in combination with cetuximab will be evaluated for antitumor activity in subjects by examining its effects on accepted clinical endpoints. Progression-free survival (PFS) will be evaluated in subjects treated with EMD 1201081 plus cetuximab compared to cetuximab alone in cetuximab-naïve subjects with R/M SCCHN who have progressed on a cytotoxic therapy.

Cetuximab, approved in colorectal cancer and SCCHN in combination with platinum-based chemotherapy and SCCHN in combination with radiotherapy in the EU, will be provided as investigational medicinal product (IMP) in this study. Commercially available Cetuximab will be provided in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent prior to any trial-specific procedure
* Male or female subjects age greater than or equal to (>=) 18 years with R/M SCCHN
* Histologically confirmed R/M SCCHN, documented in the medical record
* History of progressing disease on a first-line cytotoxic chemotherapy regimen for R/M SCCHN, such as 5-fluorouracil (FU) plus cisplatin, or taxanes. (A history of chemotherapy or radiotherapy for localized disease was not considered a first-line regimen)
* The subject is suited for systemic therapy in the opinion of the Investigator
* At least one radiographically documented lesion measurable according to response evaluation criteria in solid tumors (RECIST) 1.0. All target lesions are to be measurable (that is, the lesion must be adequately measurable in at least one dimension; longest diameter to be recorded as >= 2 centimeter (cm) by conventional techniques or >= 1 centimeter (cm) by spiral computed tomography [CT] scan). Target lesions are to be selected from the required protocol imaging. If the sole site of measurable disease is in a prior radiation field, there has to be unequivocal evidence of progression at >= 8 weeks since the completion of radiation or a positive biopsy
* Eastern cooperative oncology group performance status (ECOG PS) of 0 or 1
* If female, either post-menopausal, surgically sterile, or having a negative urine or serum pregnancy test (beta-human chorionic gonadotropin [beta-HCG]) at screening and practicing medically accepted contraception. If male, practicing contraception if the risk of conception exists. For relevant subjects, the duration of contraception should be 1 week prior to the start of therapy through 4 weeks after receipt of trial therapy
* Recovered from previous toxicities of prior cytotoxic regimen to common terminology criteria of adverse events (CTCAE) Grade 1 (with the exception of alopecia)
* Hemoglobin >= 9 gram per deciliter (g/dL) without transfusion support; no transfusion within 7 days prior to screening)
* Neutrophils >= 1.5 * 10^9 per liter
* Platelets >= 100 * 10^9 per liter
* Prothrombin time/partial thromboplastin time (PT/PTT) less than or equal to (=<) 1.5 times the upper limit of normal (ULN) for the site, unless there is therapeutic anti-coagulation
* Serum creatinine =< 1.5 times the ULN for the site
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 times the ULN for the site
* Be willing and able to comply with the protocol procedures for the duration of the trial

Exclusion Criteria:

* History of prior exposure to cetuximab or panitumumab or any other approved or investigational anti-epidermal growth factor receptor (EGFR) agents
* Undifferentiated nasopharyngeal carcinoma
* Chemotherapy, radiotherapy or any investigational agents within 4 weeks prior to first dose of study drug
* Major surgical or planned procedure within 30 days prior to first dose of trial medication (isolated biopsies are not considered major surgical procedures)
* Active malignancy other than SCCHN, non-metastatic basal cell or squamous cell carcinoma of the skin, or second primary SCCHN
* Impaired cardiac function (for example, left ventricular ejection fraction less than [<] 45 percent defined by echocardiograph or other study), history of uncontrolled serious arrhythmia, unstable angina pectoris, congestive heart failure (new york heart association [NYHA] Grade III and IV), myocardial infarction within the last 12 months prior to trial entry, or signs of pericardial effusion
* Hypertension uncontrolled by standard pharmacologic therapies
* History of diagnosed interstitial lung disease
* Subject requires systemic anti-coagulation (example, warfarin greater than [>] 10 milligram per day [mg/day])
* Pregnancy or breastfeeding
* Legal incapacity or limited legal capacity
* Significant medical or psychiatric disease which makes the trial inappropriate in the Investigator's opinion
* Any brain metastasis and/or leptomeningeal disease (known or suspected)
* Significant pre-existing immune deficiency, such as infection of human immuno-deficiency virus (HIV) (documented or known)
* Clinically significant ongoing infection
* Known hypersensitivity to the trial treatments
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer from such disease
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Breitfeld, MD, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (35):
- United States (4):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - MGH Massachusetts General Hospital, Boston, Massachusetts
  - Montefiore Medical Center Oncology, The Bronx, New York
- Belgium (4):
  - Research Site, Brussels
  - UZ Gent, Ghent
  - Research Site, Wilrijk
  - Cliniques Universitaires Mont-Godinne, Yvoir
- Czechia (4):
  - Research Site, Brno
  - Research Site, Kladno
  - Research Site, Pardubice
  - Ustav radiacni onkologie Fakultni nemacnice Na Bulovce, Prague
- France (2):
  - Research Site, Montpellier
  - Research Site, Villejuif
- Hungary (7):
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyiregyahaza
  - Szegedi Tudomayegyetem Altalanos Orvostudomanyi Kar Onkoterapias Klinika, Szeged
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Zala Megyei Kohaz Kulsokorhaz Onkologia Osztaly, Zalaegerszeg
- Poland (3):
  - SPZOZ Centrum Onkologi Liemi Lubelskiej, II Odzial Radioterapiii z pododdzialem Chemioterpii, Lublin
  - Zaklad Opleki Zdrowotnej MSWIA z Warminsko-Mazurskim Centrum Onkologil, Oddziat Chemioterapli, Olsztyn
  - Centrum Onkologi - Instytut im. Marii Sklodowskiej-Curie, Klinika Nowotworow Glowy i Szyi (NCI), Warsaw
- Slovakia (2):
  - Onkologicky ustav Sv. Alzbety, Bratislava
  - Nemocnice s poliklinikou Zilina, Žilina
- United Kingdom (9):
  - Velindre Cancer Centre, Cardiff
  - Research Site, Conventry
  - MHCW, Coventry
  - St. James' University Hospital, Leeds
  - Research Site, London
  - The Christie NHS FT, Manchester
  - Research Site, Newcastle upon Tyne
  - Weston Park Hospital, Sheffield
  - Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Result] Ruzsa A, Sen M, Evans M, Lee LW, Hideghety K, Rottey S, Klimak P, Holeckova P, Fayette J, Csoszi T, Erfan J, Forssmann U, Goddemeier T, Bexon A, Nutting C; NA EMD 1201081 Study Group. Phase 2, open-label, 1:1 randomized controlled trial exploring the efficacy of EMD 1201081 in combination with cetuximab in second-line cetuximab-naive patients with recurrent or metastatic squamous cell carcinoma of the head and neck (R/M SCCHN). Invest New Drugs. 2014 Dec;32(6):1278-84. doi: 10.1007/s10637-014-0117-2. Epub 2014 Jun 4. PMID 24894651
- See also: Related Info — http://www.cancer.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 17 Dec 2009; Last participant signed informed consent: 15 Aug 2011; Clinical data cut-off: 11 Jan 2012.
Pre-assignment Details: Of the 123 participants, 106 were randomized and 17 were screen failures (12 did not meet all eligibility criteria, 1 experienced progressive disease, 3 had unspecified reasons and data on 1 participant was missing). One participant who was not randomized but received cetuximab+EMD 1201081, was included in the safety population (107 participants).
Groups:
- Cetuximab Plus EMD 1201081: Cetuximab weekly (initial dose 400 milligram per square meter [mg/m^2] over 120 minutes followed by 250 mg/m^2 intravenous infusion over 60 minutes) and EMD 1201081 weekly (0.32 milligram per kilogram [mg/kg] by subcutaneous injection) was administered in 3-week treatment cycle until disease progression. Participants who had discontinued cetuximab due to toxicity in cetuximab monotherapy arm, continued to receive EMD 1201081 monotherapy until disease progression or participant elected to withdraw from the trial. The total treatment period was approximately 18 months.
- Cetuximab Monotherapy: Cetuximab weekly (initial dose 400 mg/m^2 over 120 minutes followed by 250 mg/m^2 intravenous infusion over 60 minutes) was administered in 3-week treatment cycle until disease progression. Participants who had discontinued cetuximab due to toxicity of cetuximab monotherapy, continued to receive EMD 1201081 monotherapy until disease progression or participant elected to withdraw from the trial. The total treatment period was approximately 18 months.
Period: Overall Study
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Started | 54 (One participant was treated with study drug 'Cetuximab Plus EMD 1201081' but was not randomized) | 53
Completed | 8 | 16
Not Completed | 46 | 37
Not completed — Adverse Event | 4 | 5
Not completed — Death | 4 | 6
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Progressive disease | 32 | 17
Not completed — Symptomatic deterioration | 2 | 5
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the randomized participants who had received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (7.03) | 56.8 (10.03) | 56.8 (8.62)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Time: Independent Read Assessments
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause within 60 days of the last tumor assessment or randomization. Participants without event were censored on the date of last tumor assessment.
Time Frame: Every 6 weeks until disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, 17 Dec 2009 until cut-off date (11 Jan 2012)
Population: ITT population included all the randomized participants who had received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Number analyzed (Participants) | 53 | 53
months | 1.5 [1.3 to 2.6] | 1.9 [1.5 to 2.9]
Statistical Analysis 1: Comparison: Cetuximab Plus EMD 1201081 vs Cetuximab Monotherapy; Test type: Superiority or Other; p = 0.793, Stratified log rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.7 to 1.6]

2. Secondary Outcome: Percentage of Participants With Objective Response: Independent Read Assessments
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) as assessed by Independent Read. As per RECIST v1.0 for target lesions and assessed by MRI: CR = Disappearance of all target lesions; PR = at least 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Every 6 weeks until disease progression, reported between day of first participant randomized, that is, 17 Dec 2009 until cut-off date (11 Jan 2012)
Population: ITT population included all the randomized participants who had received study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Number analyzed (Participants) | 53 | 53
percentage of participants | 5.7 [1.2 to 15.7] | 5.7 [1.2 to 15.7]
Statistical Analysis 1: Comparison: Cetuximab Plus EMD 1201081 vs Cetuximab Monotherapy; Test type: Superiority or Other; p > 0.999, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants With Disease Control: Independent Read Assessments
Description: Percentage of participants with disease control, defined as having achieved CR or PR or stable disease (SD) as the tumor response according to radiological assessments (based on RECIST Version 1.0 criteria), was reported. As per RECIST v1.0 for target lesions and assessed by MRI: CR = disappearance of all target lesions; PR = at least 30% decrease in the sum of the longest diameter of target lesions; SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: as for outcome 2
Population: ITT population included all the randomized participants who had received study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Number analyzed (Participants) | 53 | 53
percentage of participants | 37.7 [24.8 to 52.1] | 43.4 [29.8 to 57.7]
Statistical Analysis 1: Comparison: Cetuximab Plus EMD 1201081 vs Cetuximab Monotherapy; Test type: Superiority or Other; p = 0.557, Cochran-Mantel-Haenszel

4. Secondary Outcome: Overall Survival (OS) Time
Description: The overall survival (OS) time was defined as the time from randomization to death. Participants without event were censored at the last date known to be alive or at the clinical cut-off date, whatever was earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, that is, 17 Dec 2009 until cut-off date, (11 Jan 2012)
Population: ITT population included all the randomized participants who had received study treatment. Overall survival data was analyzed only for participants who received cetuximab plus EMD 1201081.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Number analyzed (Participants) | 53 | 0
months | 6.3 [4.2 to 9.0] |

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. A Serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Time from first dose up to Day 42 to 49 after last dose of trial treatment, reported between day of first participant randomized, that is, 17 Dec 2009 until cut-off date, (11 Jan 2012)
Population: Safety population included all the participants who received at least 1 dose study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Number analyzed (Participants) | 54 | 53
participants
  TEAEs | 52 | 53
  Serious TEAEs | 27 | 23

ADVERSE EVENTS:
Time Frame: Time from first dose up to Day 42 to 49 after last dose of trial treatment, reported between day of first participant randomized, that is, 17 Dec 2009 until cut-off date, (11 Jan 2012)
Description: An AE is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Cetuximab Plus EMD 1201081 | Cetuximab Monotherapy
Serious Adverse Events (participants affected / at risk) | 27/54 | 23/53
Other Adverse Events (participants affected / at risk) | 51/54 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus EMD 1201081 (N=54) | Cetuximab Monotherapy (N=53)
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
ADDISON'S DISEASE (Endocrine disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
TONGUE HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DEATH (General disorders) | 0 | 1
DEVICE LEAKAGE (General disorders) | 1 | 0
DISEASE PROGRESSION (General disorders) | 3 | 1
FACE OEDEMA (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1
PNEUMATOSIS (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 0
CATHETER SITE INFECTION (Infections and infestations) | 2 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
TRACHEOSTOMY MALFUNCTION (Injury, poisoning and procedural complications) | 0 | 2
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
TUMOUR NECROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
POLYNEUROPATHY (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
HAEMORRHAGE (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus EMD 1201081 (N=54) | Cetuximab Monotherapy (N=53)
ANAEMIA (Blood and lymphatic system disorders) | 9 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0
CONSTIPATION (Gastrointestinal disorders) | 8 | 4
DIARRHOEA (Gastrointestinal disorders) | 6 | 10
DYSPHAGIA (Gastrointestinal disorders) | 5 | 5
NAUSEA (Gastrointestinal disorders) | 8 | 4
STOMATITIS (Gastrointestinal disorders) | 9 | 6
VOMITING (Gastrointestinal disorders) | 7 | 3
ASTHENIA (General disorders) | 7 | 4
CHEST PAIN (General disorders) | 0 | 3
CHILLS (General disorders) | 5 | 1
FATIGUE (General disorders) | 8 | 12
INJECTION SITE ERYTHEMA (General disorders) | 3 | 0
INJECTION SITE INFLAMMATION (General disorders) | 4 | 0
INJECTION SITE PAIN (General disorders) | 3 | 0
INJECTION SITE REACTION (General disorders) | 11 | 0
PYREXIA (General disorders) | 9 | 3
BRONCHITIS (Infections and infestations) | 2 | 4
CATHETER SITE INFECTION (Infections and infestations) | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 1
PNEUMONIA (Infections and infestations) | 1 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 4
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 6
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 10 | 9
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 2
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
DIZZINESS (Nervous system disorders) | 5 | 2
HEADACHE (Nervous system disorders) | 5 | 7
ANXIETY (Psychiatric disorders) | 1 | 6
INSOMNIA (Psychiatric disorders) | 4 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 4
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
ACNE (Skin and subcutaneous tissue disorders) | 5 | 4
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 12 | 16
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 | 5
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 3
RASH (Skin and subcutaneous tissue disorders) | 16 | 18
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 6 | 3
HYPERTENSION (Vascular disorders) | 2 | 3
HYPOTENSION (Vascular disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
Few of the secondary outcome measures were planned and later removed due to Sponsor's decision to discontinue development of EMD 1201081. Overall survival data was analyzed only for participants who received EMD 1201081 plus cetuximab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less